CLINICAL TRIAL: NCT00298779
Title: An Open-Label Study to Assess the Effect of Omeprazole Administration on the Pharmacokinetics of VELCADE in Subjects With Either Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Brief Title: Open-Label Study to Assess the Effect of Omeprazole on the Pharmacokinetics of VELCADE in Patients With Either Advanced Solid Tumors or Non-Hodgkin's Lymphoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-CAN-1001; NCT00107302 (obsolete NCT alias)
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Tumors; Non-Hodgkins's Lymphoma
Keywords: patients with advanced solid tumors or Non-Hodgkins's Lymphoma
MeSH Terms: conditions — Neoplasms | interventions — Omeprazole; Bortezomib

INTERVENTIONS:
Drug: omeprazole and bortezomib

SUMMARY:
This is an open-label, randomized, multiple-dose, multicenter Pharmacokinetics drug-drug interaction study in patients with advanced solid tumors, including non-Hodgkin's lymphoma, who are in need of anti-tumor therapy. In addition, the impact of omeprazole on the pharmacodynamics of VELCADE will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:1) Male or female at least 18 y/o 2)Weigh >/= 50 kg (110lbs) and a BMI of </= 28kg/m2;3)life expectancy >/= 3 mos; 4)Karnofsky Performance Status >/=70%; 5)Women must be menopausal. 3)Men must agree to use an acceptable method of contraception for the duration of the study.4)Must sign an informed consent document indicating understanding of the purpose and procedures required for the study;5)informed consent for genetic testing 6)Subjects have advanced solid tumor (including non-Hodgkin's lymphoma).7)resolution of reversible toxicities considered related to any prior antineoplastic therapies before entry; 8)must be able to swallow capsules whole; -

Exclusion Criteria:1)Prior exposure to VELCADE.2)Has known hypersensitivity or intolerance to omeprazole, boron, mannitol or heparin. 3)Medical history of of liver or renal insufficiency; significant cardiac, vascular, pulmonary, GI, endocrine, neurologic, rheumatologic, pyschiatric or metabolic disturbances. 4)Uncontrolled diabetes. 5)history of hypotension or decreased blood pressure;6)Uncontrolled or severe cardiovascular disease incl. myocardial infarction within 6 mos of enrollment; 7)History of alcohol/drug abuse. 8)Presence of HIV antibodies, hepatitis C antibodies or hepatitis B. 9)active systemic infection requiring treatment; 10)Pregnant or breastfeeding' 11)neuropathy >/= Gr.1; 12)transfusion dependence; 12)pre-planned surgeries or procedures that would interfere with conduct of study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
The investigator will determine the patient's response to VELCADE treatment following completion of Cycle 2 (Day 21). | completion of cycle 2 - Day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Crowley Medical Research Center, Dallas, Texas, United States